CLINICAL TRIAL: NCT03951935
Title: WALK-LSS - Muscle Function and Pelvic Stability While Walking in Patients With Symptomatic Lumbar Spinal Stenosis
Brief Title: Muscle Function and Pelvic Stability While Walking in Patients With Symptomatic Lumbar Spinal Stenosis
Acronym: WALK-LSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Klinik für Radiologie und Nuklearmedizin, University Hospital Basel (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-00331; ch19Muendermann2
Record Dates: First submitted 2019-05-06; First posted 2019-05-16 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Symptomatic Lumbar Spinal Stenosis; Lumbar Spinal Stenosis
Keywords: pelvic stability; lumbo- pelvic- hip complex; lumbo-pelvic-hip muscles
MeSH Terms: conditions — Spinal Stenosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sLSS: patients diagnosed with sLSS scheduled for decompression surgery
  Interventions: Other: Oswestry Disability Index (ODI) questionnaire; Diagnostic Test: self-paced walking test (SPWT)
- control subjects: healthy, age-matched control subjects
  Interventions: Other: Oswestry Disability Index (ODI) questionnaire; Diagnostic Test: self-paced walking test (SPWT)

INTERVENTIONS:
Other: Oswestry Disability Index (ODI) questionnaire — Participant's level of low back pain and the extent to which the pain impacts his/ her daily life activities and social life are estimated with the standardized Oswestry Disability Index questionnaire
Diagnostic Test: self-paced walking test (SPWT) — walking back and forth at a self-selected pace along a hallway at the University Hospital until the onset of claudication, pain or until reaching the time limit of 30 minutes. Kinematic and electromyographic (EMG) data will be recorded every 3 minutes.

SUMMARY:
This study is to quantify changes in muscle activity and pelvic stability during prolonged walking in patients with symptomatic lumbar spinal stenosis (sLSS) and healthy control subjects and to determine their association with the severity of the stenosis and the crosssectional area and fatty atrophy of lumbo-pelvic-hip muscles.

ELIGIBILITY:
Inclusion Criteria patients:

* Diagnosed symptomatic lumbar spinal stenosis
* Availability of lumbar MR images
* Scheduled for decompressive surgery at the University Hospital Basel

Exclusion Criteria patients:

* Prior decompressive surgery
* Body Mass Index (BMI) ≥ 35 kg/m2
* Additional pathologies that influence the mobility of the pelvis
* Use of walking aids
* Inability to provide informed consent

Exclusion Criteria healthy control subjects:

* BMI ≥ 35 kg/m2
* Pain in the lower extremity or lower back in the previous 6 months
* Prior surgery of the lumbo-pelvic-hip complex
* History of claudications
* Neurological or orthopaedic conditions that may influence gait
* Inability to provide informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 20 patients diagnosed with sLSS scheduled for decompression surgery at the University Hospital Basel
  * 20 healthy, age-matched control subjects
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) questionnaire | the day before decompression surgery
  Participant's level of low back pain and the extent to which the pain impacts his/ her daily life activities and social life; ten self-administered items compiling the ODI are: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life, travelling. The resulting scores are presented as scores from 0 (no impact) to 100 (bed bound and extremely limited). Higher values represent a worse outcome.
Muscle activation assessed by Electromyography (EMG) | scheduled the day before decompression surgery
  Muscle activation of the multifidus, gluteus medius, erector spinae (longissimus), transversus abdominis muscles will be measured bilaterally using a 12- channel EMG system (myon AG, Schwarzenberg, Switzerland). Surface electrodes will be placed on these muscles (sampling rate = 2000 Hz). For each muscle, the frequency spectrum will be computed for each recording. Muscle fatigue will be defined as the slope of the mean frequency during the self-paced walking test (SPWT)
Pelvic stability | the day before decompression surgery
  Pelvic stability will be assessed using an inertial sensor-based gait analysis system, more precisely by the sensor attached to the posterior superior iliac spine (RehaGait, Hasomed GmbH, Magdeburg, Germany). Pelvic stability will be measured in three planes (sagittal, transversal, frontal). Each sensor comprises a 3-axis accelerometer (± 16 g), a 3-axisgyroscope (± 2000 °/s) and a 3-axis compass (± 1.3 Gs). Dynamic stability will be defined as the root mean square ratio of the pelvic acceleration in each direction (anteroposterior, medio-lateral, vertical) normalized to walking Speed.
Cross-sectional area (CSA) of lumbo-pelvic-hip muscles | the day before decompression surgery
  Quantitative measurements of the CSA will be obtained from an axial T1 vibe Dixon transversal sequence and will be assessed by using an imaging software (syngo.via, Siemens Healthineers, Erlangen, Germany). The Dixon method represents a commonly used method to suppress the signal of fat in magnetic resonance imaging (MRI). The range of interest (ROI) will be defined manually on L3/L4- and on L4/L5-level and will include the CSA of the musculus (m.) erector spinae and the m. psoas major bilaterally. The CSA will be set in relation to the subject's Body mass. MRIs are routinely acquired in patients as diagnostics prior to surgery. The T1 vibe Dixon transversal sequence is not part of the standardized imaging protocol and will be added to the protocol for eligible patients for the purpose of this study.
Fatty atrophy of lumbo-pelvic-hip muscles | the day before decompression surgery
  The fatty atrophy of the lumbo-pelvic-hip muscles will be assessed with an axial T2-weighted sequence enabling determining the fat fraction. The ROI will be defined manually on L3/L4- and on L4/L5-level and will include the erector spinae and the psoas major bilaterally. This sequence is part of the standardized imaging protocol.
walking capacity assessed by self-paced walking test distance (SPWT) | the day before decompression surgery
  The SPWT will be conducted on a level surface in a hallway at the University Hospital. The duration, measured with a stopwatch by the administrator, and pain scores during walking, ranked between 0 and 10 and given every 5 minutes via oral feedback by the participant, will be assessed.
Grading of Severity of Lumbar Spinal Stenosis using the classification by Schizas | the day before decompression surgery
  The stenosis grade will be assessed using the classification by Schizas.The 4-grade based classification is based on the morphology of the dural sac as observed on T2 axial MRI based on the rootlet/ cerebrospinal fluid ratio. Grade A stenosis: there is clearly cerebrospinal fluid (CSF) visible inside the dural sac, but its distribution is inhomogeneous.
  Grade B stenosis: the rootlets occupy the whole of the dural sac, but they can still be individualized. Some CSF is still present.
  Grade C stenosis: no rootlets can be recognized, the dural sac demonstrating a homogeneous gray signal with no CSF signal visible. There is epidural fat present posteriorly.
  Grade D stenosis: in addition to no rootlets being recognizable there is no epidural fat posteriorly. Grade A is defined as no or minor stenosis, B as moderate stenosis, C as severe stenosis, and D as extreme stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, Prof. Dr. MD, Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland